CLINICAL TRIAL: NCT06923540
Title: Evaluating the Impact of IV Acetaminophen on Opioid Consumption in the Postoperative Period in Patients Undergoing Abdominal Surgery
Brief Title: Intravenous Acetaminophen to Reduce Post-operative Opioid Consumption
Acronym: ACETAPOP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-12623
Record Dates: First submitted 2025-03-13; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Analgesia; Opioid Consumption, Postoperative; Acetaminophen; Abdominal Surgeries; Post Operative Bowel Dysfunction; Post Operative Nausea and Vomiting; Post Operative Pain Control; Mobility; Epidural Analgesia; Length of Stay; Pain Management
Keywords: IV acetaminophen; intravenous acetaminophen; acetaminophen; post operative analgesia; nil per os; npo; post operative pain; opioid consumption; abdominal surgery; hepato-biliary surgery; digestive surgery; pancreatic surgery; gynecologic surgery; post operative nausea and vomiting; post operative mobility; hospitalization length of stay; co-analgesia
MeSH Terms: conditions — Vomiting; Agnosia; Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: The study design is quasi-experimental in pre post fashion.
  * Part 1: participants will receive the standard post-operative protocol, which includes Acetaminophen PO or IR.
  * Part 2 : participants will receive the modified post-operative protocol, which includes IV Acetaminophen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-intervention arm (standard protocol containing PO or IR Acetaminophen) (No Intervention): This arm will receive the protocol currently used at the CHUM surgical units for post operative pain management, which includes PO or IR acetaminophen.
- Post-intervention arm (modified protocol containing IV Acetaminophen) (Active Comparator): This arm will receive a modified protocol version of the one used at the CHUM surgical units for post operative pain management, which includes IV acetaminophen.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — This intervention will be administered to patients undergoing abdominal surgery who are nil per os (NPO) directly after surgery. This patient group has not been properly studied in other clinical studies using IV Acetaminophen. The study aim is to determine if patients who have an altered enteral route may benefit from IV Acetaminophen.
  Arms: Post-intervention arm (modified protocol containing IV Acetaminophen)

SUMMARY:
Acetaminophen (Tylenol) is a commonly used medication after surgery to control pain. Tablets for oral use and suppositories for rectal use are the most frequently employed forms of acetaminophen after surgery. Intravenous (IV) acetaminophen is widely used in several countries but is not a standard medication for the adult population in Canada. It is mainly considered when it is impossible to take medication in tablet or suppository form. Opioids (Morphine, Hydromorphone, Oxycodone, etc.) are another class of medications commonly used after surgery for pain management. While they are generally very effective and stronger than acetaminophen or other pain relievers (e.g., ibuprofen/Advil), reducing their use is preferable, as they can cause various side effects such as nausea, dizziness, and dependence. IV acetaminophen may help control pain while also reducing opioid consumption. However, there are few high-quality scientific studies proving the benefits of IV acetaminophen compared to other forms, such as tablets or suppositories. Acetaminophen has been available in Canada for many years and has already been recommended for use in Quebec by the Institut national d'excellence en santé et services sociaux (INESSS) under certain conditions. This study aims to validate its benefits with clear data.

DETAILED DESCRIPTION:
In 2019, the Institut national d'excellence en santé et services sociaux (INESSS) stated that IV acetaminophen is an acceptable short-term pain treatment option in combination with opioid analgesics for adults and children aged two years and older when oral (PO) and rectal (IR) acetaminophen cannot be used. Despite this recommendation, there is limited data on IV acetaminophen in patients with a compromised enteral route, even though this is likely one of the populations that could benefit the most from such an intervention. Patients undergoing abdominal surgeries are a prominent example of individuals with a compromised enteral route. Some data exist for other types of surgeries, such as orthopedic surgery. However, such data is challenging to extrapolate to abdominal surgeries since orthopedic surgery does not affect the digestive system. Furthermore, several studies use comparators that do not accurately reflect clinical practice, such as placebo. This study will therefore use standard treatment as a comparator, allowing for a better assessment of IV acetaminophen's role in the therapeutic arsenal.

IV acetaminophen is approved and marketed in Canada. It is not an investigational product. Furthermore, it is currently used in other hospital centers and has already been used at the Centre hospitalier de l'Université de Montréal (CHUM). Given current budgetary limitations, PO and IR formulations of acetaminophen have been preferred over the IV formulation, as their economic burden is less than IV acetaminophen.

Currently, pharmacists play a central role in the healthcare system as medication experts and key players in patient care in both community and hospital settings. Over the years, pharmacists in Québec have also become prescribers by law. They are valuable allies in hospitals, ensuring proper treatment follow-up and continuously validating that pharmacological care standards for patients of the CHUM are met.

The research question is as follows: Compared to standard local postoperative treatment, does IV acetaminophen reduce the amount of opioids administered within the first 72 postoperative hours in patients with a compromised enteral route in the abdominal surgery units of a Québec university hospital center?

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Underwent abdominal surgery
* Underwent elective surgery.
* Hospitalized in the digestive surgery, hepatobiliary and pancreatic surgery, or gynecology and gynecologic oncology units at CHUM.
* Declared NPO immediately post-surgery, meaning they cannot take oral medications.

Exclusion Criteria:

* Hypersensitivity to acetaminophen or an excipient in the administered formulations
* Hepatic insufficiency with a Child-Turcotte-Pugh score of B or C.
* Weight < 50 kg (patients requiring a lower acetaminophen dose).
* Active pregnancy or breastfeeding.
* Opioid use disorder (OUD) under active treatment
* Non-opioid-naïve patients: those who received a long-acting opioid within seven days preceding surgery. This criterion will be verified through patient interviews and cross-checked with medical records.
* Use of illicit recreational substances.
* Prior participation in this study.
* Ectopic patients: physically located in a unit other than digestive surgery (11 South), hepatobiliary and pancreatic surgery (14 South), or gynecology and gynecologic oncology (12 South).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption in oral morphine milligram equivalents (MME) | 72 hours
  To determine whether the systematic use of IV acetaminophen in adult NPO patients in the postoperative context of abdominal surgery (post-intervention) reduces the average opioid consumption in oral morphine milligram equivalents (MME) over 72 hours compared to the standard protocol, which includes PO or IR acetaminophen (pre-intervention).

SECONDARY OUTCOMES:
Opioid consumption (converted to MME) at 24 and 48 hours postoperatively | 48 hours
  To determine whether the systematic use of IV acetaminophen reduces the average opioid consumption in MME over the first 24 and 48 postoperative hours in the post-intervention period compared to the pre-intervention period.

OTHER OUTCOMES:
Pain level at rest (on a scale from 0 to 10) during the first 72 hours. | 72 hours
  Compare the variation in resting pain levels during the periods of 0 to 24 hours, 24 to 48 hours, 0 to 48 hours, 48 to 72 hours, and 0 to 72 hours between the pre-intervention and post-intervention periods. This simple scale asks patients to rate their pain on a scale from zero (no pain) to ten (maximum pain).
Pain level during mobilization (on a scale from 0 to 10) during the first 72 hours | 72 hours
  Compare the average pain level during mobilization (upon standing) on postoperative days 0, 1, and 2 between the pre-intervention and post-intervention periods. This simple scale asks patients to rate their pain on a scale from zero (no pain) to ten (maximum pain)
Length of hospital stay | From date of the abdominal surgery until the date of hospital discharge, assessed up to 6 months
  Compare the length of hospital stay in days from the end of surgery until hospital discharge between the pre-intervention and post-intervention periods.
Nausea and constipation (antiemetic doses, laxative use) | 72 hours
  Compare the frequency of nausea and constipation between the pre-intervention and post-intervention periods
Functionality: time to first mobilization, mean chair time on postoperative days 1 and 2, time to return of oral intake, time to epidural discontinuation. | 72 hours
  Compare the average time (in days) before the return of an uncompromised enteral route, complete epidural weaning, and first mobilization (first time standing up) between the pre-intervention and post-intervention periods.
  Compare the average time spent seated in a chair on postoperative days 1 and 2 between the pre-intervention and post-intervention periods.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Vandenbroucke-Menu, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No